CLINICAL TRIAL: NCT06461936
Title: Intra-Tumoral Vascular Growth Patterns is a Robust Indicator of Adjuvant PD-1 Inhibitors Following Liver Resection in Hepatocellular Carcinoma: A Multicenter Cohort and Multiomics Study
Brief Title: Intra-Tumoral Vascular Growth Patterns is a Robust Indicator of Adjuvant Therapy Following Liver Resection in HCC
Status: Active, not recruiting | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: PrecisionAT
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: HCC; Adjuvant Therapy; Immunotherapy; Recurrence
MeSH Terms: conditions — Recurrence | interventions — sintilimab; lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Transcriptome, protein and metabolome sequencing were performed on frozen and paraffin-block tissues from selected patients. Paraffin-block tissues were used for spatial transcriptome analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active Surveillance Group（AC）: Patients in AC group received no adjuvant therapy after liver resection.
- Adjuvant sintilimab group（AS）: Patients in AS group received adjuvant sintilimab after liver resection.
  Interventions: Drug: Sintilimab
- Adjuvant sintilimab plus Lenvatinib group （ASL）: Patients in ASL group received adjuvant sintilimab plus lenvatinib therapy after liver resection.
  Interventions: Drug: Sintilimab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Sintilimab — Patient receives first adjuvant PD-1monoclonal antibody 2-4 weeks postoperatively, 200mg IV over 21 days for 9 cycles.
  Groups: Adjuvant sintilimab group（AS）; Adjuvant sintilimab plus Lenvatinib group （ASL）
Drug: Lenvatinib — Lenvatinib is initiated orally 2-4 weeks postoperatively for about 6 months.
  Groups: Adjuvant sintilimab plus Lenvatinib group （ASL）

SUMMARY:
Vessels that encapsulate tumor clusters (VETC) is an invasive metastatic factor in HCC independent of the epithelial mesenchyme transition (EMT), and VETC positive patients have a higher rate of postoperative recurrence. However, it is not clear how the surgical prognosis of VETC-positive patients can be improved.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common malignancy worldwide, with the number of new cases and deaths increasing yearly. Curative surgery continues to be the preferred treatment for early-stage HCC. However, some early-stage HCC often experience early recurrence after surgery, and one of the most common risk factors is microvascular invasion (MVI). Nevertheless, the overall prognosis of some MVI-negative patients is also not satisfactory. Whether there are other hidden robust risk factors for recurrence is of intense interest to clinical scientists.

In contrast to the classic capillary pattern, cobweb-like pattern of vascular is present in renal cell carcinoma, thyroid follicular carcinoma and HCC. Specifically, this particular vascular pattern is a continuous lining of sinusoid-like vessels that isolate and encapsulate individual tumor clusters, and Fang et al. named it vessels that encapsulate tumor clusters (VETC). CD34 or CD31 immunohistochemical staining of tumor tissue can easily identify the vascular pattern of VETC, which can exist at any stage of HCC, accounting for about 40%-50.6%. VETC could directly invade adjacent vascular and migrate as tumor clusters instead of epithelial-mesenchymal transition pathway, which may well explain why VETC-positive HCC is closely associated with higher postoperative recurrence rate and poor prognosis. Due to the high proportion of VETC vascular patterns and poor prognosis, it is necessary to adopt effective adjuvant treatment. Zhuan et al found that unresectable VETC+HCC could benefit from treatment with sorafenib in a subsequent study. Similarly, another study found that FGF 2 and FGFR 3-4 (rather than VEGF-A or VEGFR 1-3) were high expression in VETC+ HCC, which raise the possibility that lenvatinib is a potentially effective treatment modality. Recently, a multicenter randomized controlled trial of postoperative adjuvant Sintilimab reported encouraging positive results, suggesting the possibility of its application in VETC-positive patients. Whether the combination of lenvatinib and Sintilimab can further improve the prognosis is also worth exploring.

To address these clinical challenges, the investigators conducted a multicenter study involving three surgical cohorts with postoperative active surveillance cohort(AC), adjuvant Sintilimab cohort(AS), and adjuvant Sintilimab plus Lenvatinib cohort(ASL). The cases in the AS cohort were mainly from a previous prospective cohort study initiated by the investigator's center and a later cohort expansion (NCT05307926). Moreover, multi-omics sequencing analysis aims to further explore the molecular biological characteristics between VETC positive and negative HCC.

ELIGIBILITY:
Inclusion Criteria:

* Underwent radical hepatectomy
* No preoperative treatment
* Pathological confirmed HCC
* High-risk recurrent HCC
* Not receiving any adjuvant therapy or receiving adjuvant therapy with PD-1 monotherapy or receiving adjuvant therapy with PD-1 monotherapy in combination with Lenvatinib after surgery
* Evaluable wax block tissue as well as complete clinical information

Exclusion Criteria:

* Distant metastasis
* No available wax blocks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three cohort cases were retrospectively collected from 4 medical centers according to the study design. Most of the data of AS cohort were obtained from a prospective cohort study of Tongji Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease -free survival | From date of surgery to the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months.
  Disease-free survival was defined as the time from surgery to diagnosis of recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall survival | From date of surgery to the date of death from any cause, assessed up to 60 months.
  Overall survival was defined as the time from surgery to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes